CLINICAL TRIAL: NCT00453154
Title: Combination Chemotherapy With or Without Maintenance Sunitinib Malate (NSC 736511) for Untreated Extensive Stage Small Cell Lung Cancer: A Phase IB/Randomized Phase II Study
Brief Title: Cisplatin or Carboplatin, and Etoposide With or Without Sunitinib Malate in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00465; NCI-2009-00465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000538229; CALGB 30504 (Other: Alliance for Clinical Trials in Oncology); CALGB-30504 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Recurrent Lung Small Cell Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (Combination Chemotherapy + Sunitinib Maintenance) (Experimental): Participants will receive the following combination chemotherapy for 4-6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle OR Carboplatin AUC = 5* by IV Etoposide 100 mg/m^2 by IV over 1 hour on days 1, 2, and 3 every cycle
  Maintenance: Following 4-6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Sunitinib Malate
- Arm II (Combination Chemotherapy + Placebo Maintenance) (Active Comparator): Participants will receive the following combination chemotherapy for 4-6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle OR Carboplatin AUC = 5* by IV Etoposide 100 mg/m2 by IV over 1 hour on days 1, 2, and 3 every cycle
  Maintenance: Following 4-6 cycles of combination chemotherapy, start placebo at 150 mg on day 1, then 37.5 daily until disease progression.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Other: Placebo Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (Combination Chemotherapy + Placebo Maintenance)
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
  Arms: Arm I (Combination Chemotherapy + Sunitinib Maintenance)

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of sunitinib malate and to see how well it works when given together with cisplatin or carboplatin and etoposide in treating patients with extensive-stage small cell lung cancer. Drugs used in chemotherapy, such as cisplatin, carboplatin, and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether cisplatin or carboplatin and etoposide are more effective when given with or without sunitinib malate in treating small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the phase II dose for sunitinib (sunitinib malate) combined with cisplatin and etoposide. (Phase IB) II. To compare the progression-free survival of patients with extensive stage small cell lung cancer treated with cisplatin or carboplatin and etoposide followed by maintenance sunitinib to patients receiving the same chemotherapy followed by placebo. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the single agent response rate for sunitinib given as monotherapy after chemotherapy. (Phase II) II. To assess the overall survival of patients treated with cisplatin or carboplatin and etoposide followed by sunitinib. (Phase II) III. To evaluate the toxicity and tolerability of maintenance sunitinib after cisplatin or carboplatin and etoposide. (Phase II) IV. To determine the association between vascular endothelial growth factor (VEGF) plasma levels and tumor response. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of sunitinib malate followed by a randomized phase II study.

PHASE I (close to accrual 5/17/08):

COMBINATION THERAPY: Patients receive cisplatin or carboplatin intravenously (IV) on day 1, etoposide IV on days 1-3, and sunitinib malate orally (PO) once daily (QD) on days 1-14. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive sunitinib malate PO alone QD. Treatment continues in the absence of disease progression or unacceptable toxicity.

PHASE II:

COMBINATION THERAPY: Patients receive cisplatin or carboplatin and etoposide as in Phase I. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Beginning 3-8 weeks after completion of combination chemotherapy or >= 4 courses of combination therapy, patients with a responding or stable disease are randomized to 1 of 2 treatment arms. All patients must be euthyroid before starting on maintenance therapy.

ARM I: Patients receive sunitinib malate PO QD. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with disease progression may cross over to Arm I.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically documented small cell lung cancer

  * Eligible disease stages: the extensive disease classification for this protocol includes all patients with disease sites not defined as limited stage; limited stage disease category includes patients with disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal, and/or ipsilateral supraclavicular nodes; extensive stage patients are defined as those patients with extrathoracic metastatic, malignant pleural effusion, bilateral or contralateral supraclavicular adenopathy or contralateral hilar adenopathy
* All patients must have measurable disease:

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
  * Lesions that are considered non-measurable, which would make the patient not eligible, include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No prior chemotherapy for small cell lung cancer (SCLC)
* Radiation therapy must have been completed at least one week before initiation of protocol therapy
* Common Toxicity Criteria (CTC) performance status:

  * Phase IB: 0-1
  * Phase II: 0-2
* No "currently active" second malignancy other than non-melanoma skin cancers
* No history of brain metastases, spinal cord compression, or carcinomatous meningitis
* No ongoing cardiac dysrhythmias, atrial fibrillation, or QTc interval >= 500 msec; the use of agents with proarrhythmic potential (e.g., quinidine, procainamide, disopyramide, sotalol, probucol, pedridel, haloperidol, risperidone, indapamide, flecainide) is not recommended while on protocol therapy
* Patients with class I New York Heart Association (NYHA) are eligible; patients with a history of class II NYHA are eligible, provided they meet the following criteria:

  * Patients with a history of class II heart failure who are asymptomatic on treatment
  * Patients with prior anthracycline exposure
  * Patients who have received central thoracic radiation that included the heart in the radiotherapy port
* Patients with a history of class III or IV NYHA heart failure within 12 months prior to registration are not eligible
* Additionally, no myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft or stenting, cerebrovascular accident including transient ischemic attack, or pulmonary embolism within the last year
* Patients with hypertension that cannot be controlled by medications (> 150/100 mmHg despite optimal medical therapy) are not eligible
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; Note: Low molecular weight heparin is permitted provided the patient's prothrombin time (PT) international normalized ratio (INR) is =< 1.5
* No evidence of hemoptysis within 4 weeks prior to starting study treatment; patients with blood-tinged or blood streaked sputum will be permitted on study if the hemoptysis amounts to less than 5 mL of blood per episode and less than 10 mL of blood per 24-hour period in the best estimate of the investigator
* None of the following within 28 days of treatment: abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, serious or non-healing wound, ulcer, or bone fracture
* The use of the following specific inhibitors and inducers of cytochrome p450, family 3, subfamily A, polypeptide 4 (CYP3A4) is not permitted; the following inhibitors of CYP3A4 are prohibited within 7 days before and during treatment with sunitinib: azole antifungals (ketoconazole, itraconazole), diltiazem, clarithromycin, erythromycin, verapamil, delavirdine, and human immunodeficiency virus (HIV) protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir); the following inducers of CYP3A4 are prohibited within 12 days before beginning and during treatment with sunitinib: rifampin, rifabutin, carbamazepine, phenobarbital, phenytoin, St. John's Wort, efavirenz, tipranavir

  * Other inhibitors and inducers of CYP3A4 may be used if necessary, but there use is discouraged
* Non-pregnant and non-nursing
* Granulocytes >= 1,500/ul
* Platelets >= 100,000/ul
* Creatinine clearance >= 70 ml/min
* Total bilirubin =< 1.5 mg/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) (patients w/ liver metastases may have AST/ALT =< 5 x ULN)
* Partial thromboplastin time (PTT) =< 1.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-03-15 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2015-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal E Ready, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (125):
- United States (125):
  - Arroyo Grande Community, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lakeland Hospital Niles, Niles, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Ventz S, Khozin S, Louv B, Sands J, Wen PY, Rahman R, Comment L, Alexander BM, Trippa L. The design and evaluation of hybrid controlled trials that leverage external data and randomization. Nat Commun. 2022 Oct 2;13(1):5783. doi: 10.1038/s41467-022-33192-1. PMID 36184621
- [Derived] Ready NE, Pang HH, Gu L, Otterson GA, Thomas SP, Miller AA, Baggstrom M, Masters GA, Graziano SL, Crawford J, Bogart J, Vokes EE. Chemotherapy With or Without Maintenance Sunitinib for Untreated Extensive-Stage Small-Cell Lung Cancer: A Randomized, Double-Blind, Placebo-Controlled Phase II Study-CALGB 30504 (Alliance). J Clin Oncol. 2015 May 20;33(15):1660-5. doi: 10.1200/JCO.2014.57.3105. Epub 2015 Mar 2. PMID 25732163
- See also: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2007 and December 2011, 156 participants were recruited.
Groups:
- Phase 1B: Participants will receive the following combination chemotherapy for 6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle Etoposide 100 mg/m^2 by IV over 1 hour on days 1, 2, and 3 every cycle Sunitinib 25 mg oral, daily days 1-14 every cycle
  Maintenance: Following 6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
- Phase II Combination Chemotherapy: Participants will receive the following combination chemotherapy for 4-6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle OR Carboplatin AUC = 5* by IV Etoposide 100 mg/m^2 by IVover 1 hour on days 1, 2, and 3 every cycle
- Double Blind Placebo Maintenance With Optional Crossover: Maintenance: Following 4-6 cycles of combination chemotherapy, start placebo at 150 mg on day 1, then 37.5 daily until disease progression.
  At progression, participants receiving placebo could cross over to receive open label sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
- Double Blind Sunitinib Maintenance: Following 4-6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
Period: Combination Chemotherapy
Arm/Group | Phase 1B | Phase II Combination Chemotherapy | Double Blind Placebo Maintenance With Optional Crossover | Double Blind Sunitinib Maintenance
Started | 12 | 144 | 0 | 0
Completed | 12 | 95 | 0 | 0
Not Completed | 0 | 49 | 0 | 0
Period: Double BIind Maintenance
Arm/Group | Phase 1B | Phase II Combination Chemotherapy | Double Blind Placebo Maintenance With Optional Crossover | Double Blind Sunitinib Maintenance
Started | 0 | 0 | 46 | 49
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 46 | 49
Not completed — Adverse Event | 0 | 0 | 3 | 12
Not completed — Death | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 4
Not completed — Progression | 0 | 0 | 29 | 26
Not completed — Medical Issues | 0 | 0 | 3 | 1
Not completed — Randomized, did not receive therapy | 0 | 0 | 5 | 5
Period: Open Label Sunitinib Crossover
Arm/Group | Phase 1B | Phase II Combination Chemotherapy | Double Blind Placebo Maintenance With Optional Crossover | Double Blind Sunitinib Maintenance
Started | 0 | 0 | 18 | 0
Completed | 0 | 0 | 18 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol, participants who were randomized and received treatment were analyzed.
Groups:
- Phase I: Participants will receive the following combination chemotherapy for 6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle Etoposide 100 mg/m^2 by IV over 1 hour on days 1, 2, and 3 every cycle Sunitinib 25 mg oral, daily days 1-14 every cycle
  Maintenance: Following 6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
- Total: Total of all reporting groups
Arm/Group | Phase I | Arm I (Combination Chemotherapy + Sunitinib Maintenance) | Arm II (Combination Chemotherapy + Placebo Maintenance) | Total
Number analyzed (Participants) | 12 | 44 | 41 | 97
Age, Continuous [Median (Full Range); unit: years] | 57 [43 to 72] | 60 [39 to 69] | 61 [56 to 77] | 60 [39 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 26 | 21 | 51
  Male | 8 | 18 | 20 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 4
  White | 12 | 41 | 40 | 93
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 44 | 41 | 97
Chemotherapy Agent [Number; unit: participants] — Type of treatment received prior to maintenance randomization.
  participants
    Cisplatin | NA — Stratification factor for Phase II, not collected for Phase I patients. | 12 | 11 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Carboplatin | NA — Stratification factor for Phase II, not collected for Phase I patients. | 32 | 30 | NA — Total not calculated because data are not available (NA) in one or more arms.
Number of combination chemotherapy cycles [Number; unit: participants] — Number of cycles of combination chemotherapy received prior to maintenance randomization.
  participants
    < 6 cycles | NA — Stratification factor for Phase II, not collected for Phase I patients. | 12 | 9 | NA — Total not calculated because data are not available (NA) in one or more arms.
    6 cycles | NA — Stratification factor for Phase II, not collected for Phase I patients. | 32 | 32 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated of Sunitinib Combined With Cisplatin and Etoposide (Phase I)
Description: The maximum tolerated dose is defined at the highest sunitinib dose at which less than one third of participants develop a dose limiting toxicity (DLT). A DLT is defined as: delay of beginning cycle 2 of chemotherapy by > 7 days due to neutropenia, grade 4 hematologic toxicity lasting greater than 1 week (chemotherapy alone would be expected to cause significant grade 4 hematologic toxicity) or grade 3 or 4 nonhematologic toxicity (excluding grade 3 or 4 fatigue if the patient is found to be hypothyroid and responds to fatigue < grade 3 with thyroid replacement therapy).
Time Frame: 21 days
Population: Due to safety concerns, the study committee discontinued sunitinib from combination chemotherapy to study single agent sunitinib in the maintenance setting.
Measure: Number; unit: mg/day
Groups:
- Cohort 1: Participants will receive the following combination chemotherapy for 6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle Etoposide 100 mg/m^2 by IV over 1 hour on days 1, 2, and 3 every cycle Sunitinib 25 mg oral, daily days 1-14 every cycle
  Maintenance: Following 6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
- Cohort 2: Participants will receive the following combination chemotherapy for 6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle Etoposide 100 mg/m^2 by IV over 1 hour on days 1, 2, and 3 every cycle Sunitinib 37.5 mg oral, daily days 1-14 every cycle
  Maintenance: Following 6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
- Cohort 3: Participants will receive the following combination chemotherapy for 6 cycles (21 days):
  Cisplatin 80 mg/m^2 by IV over 1 hour on day 1 every cycle Etoposide 100 mg/m^2 by IV over 1 hour on days 1, 2, and 3 every cycle Sunitinib 50 mg oral, daily days 1-14 every cycle
  Maintenance: Following 6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 12 | 0 | 0
mg/day | 25 |  |

2. Primary Outcome: Progression-free Survival (Phase II)
Description: Progression free survival (PFS) was defined as the time from maintenance randomization to progression or death of any cause. Progression free and alive patients were censored at the date of last follow-up. The median PFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 3 years
Population: Participants who were randomized to maintenance were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Combination Chemotherapy + Sunitinib Maintenance) | Arm II (Combination Chemotherapy + Placebo Maintenance)
Number analyzed (Participants) | 44 | 41
months | 3.7 [1.8 to 4.3] | 2.1 [1.6 to 2.6]
Statistical Analysis 1: Comparison: Arm I (Combination Chemotherapy + Sunitinib Maintenance) vs Arm II (Combination Chemotherapy + Placebo Maintenance); Test type: Non-Inferiority or Equivalence — Using a 1-sided significance level of 0.15, the study has approximately 89% power to reject the null hypothesis; p = 0.02, Log Rank — All randomization was done using a permuted-block scheme with a block size of 6, stratified by combination chemotherapy (cisplatin vs carboplatin) and number of combination chemotherapy cycles (< 6 vs 6 cycles); Hazard Ratio (HR) = 1.62, 70% CI 2-sided [1.27 to 2.08]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to 3 years
Population: Participants who were randomized to maintenance were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Combination Chemotherapy + Sunitinib Maintenance) | Arm II (Combination Chemotherapy + Placebo Maintenance)
Number analyzed (Participants) | 44 | 41
months | 9.0 [8.0 to 12.7] | 6.9 [5.4 to 11.8]

4. Secondary Outcome: Number of Participants With Overall Tumor Response
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): disappearance of all target lesions; Partial Response (PR) 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria. Overall tumor response is the total number of CR and PRs.
Time Frame: Up to 3 years
Population: Participants who were randomized to maintenance were analyzed.
Measure: Number; unit: participants
Arm/Group | Arm I (Combination Chemotherapy + Sunitinib Maintenance) | Arm II (Combination Chemotherapy + Placebo Maintenance)
Number analyzed (Participants) | 44 | 41
participants
  Complete Response | 3 | 0
  Partial Response | 4 | 5

5. Other Pre Specified Outcome: Change in Plasma Levels of VEGF Prior to, During Single-agent, and Following Treatment With Sunitinib Malate
Description: The frequency of tumor response by the optimally dichotomized VEGF levels will be tabulated and their association will be tested by Fisher's exact test as well as the maximally selected rank test. The association of the VEGF levels as continuous predictor with tumor response will be tested by Wilcoxon rank sum test. Further assessments of the association of the VEGF levels as> continuous or binary variables and the tumor response will be implemented in a logistic regression while adjusting for other covariates such as performance status, weight loss and age
Time Frame: Baseline to within 7 days of sunitinib/placebo therapy discontinuation
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Plasma Levels of PDGF
Description: Correlated with clinical outcome (response and survival).
Time Frame: Baseline to within 7 days of sunitinib/placebo therapy discontinuation
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 84 participants were evaluable for adverse events.
Groups:
- Arm I (Combination Chemotherapy + Sunitinib Maintenance): Maintenance: Following 4-6 cycles of combination chemotherapy, start sunitinib at 150 mg on day 1, then 37.5 daily until disease progression.
- Arm II (Combination Chemotherapy + Placebo Maintenance): Maintenance: Following 4-6 cycles of combination chemotherapy, start placebo at 150 mg on day 1, then 37.5 daily until disease progression.
Arm/Group | Arm I (Combination Chemotherapy + Sunitinib Maintenance) | Arm II (Combination Chemotherapy + Placebo Maintenance)
Serious Adverse Events (participants affected / at risk) | 12/43 | 9/41
Other Adverse Events (participants affected / at risk) | 41/43 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Combination Chemotherapy + Sunitinib Maintenance) (N=43) | Arm II (Combination Chemotherapy + Placebo Maintenance) (N=41)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pancreatic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (8) | 5 (7)
Fever (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
ADH abnormal (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 5 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 6 (6) | 1 (1)
Weight loss (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Combination Chemotherapy + Sunitinib Maintenance) (N=43) | Arm II (Combination Chemotherapy + Placebo Maintenance) (N=41)
Hemoglobin decreased (Blood and lymphatic system disorders) | 22 (59) | 28 (78)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (5)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 4 (5)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 6 (18) | 2 (5)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 2 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 7 (8)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (9) | 10 (13)
Diarrhea (Gastrointestinal disorders) | 21 (41) | 13 (24)
Dry mouth (Gastrointestinal disorders) | 3 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 8 (11) | 1 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (34) | 20 (39)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 8 (13)
Chest pain (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 4 (4) | 2 (4)
Edema limbs (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 30 (91) | 31 (86)
Fever (General disorders) | 3 (3) | 2 (3)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 1 (2)
Localized edema (General disorders) | 1 (4) | 3 (3)
Pain (General disorders) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3)
Sinusitis (Infections and infestations) | 3 (8) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative respiratory injury - Trachea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (19) | 6 (26)
Alkaline phosphatase increased (Investigations) | 10 (14) | 5 (8)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (20) | 8 (16)
Blood bilirubin increased (Investigations) | 1 (6) | 0 (0)
Creatinine increased (Investigations) | 4 (19) | 2 (3)
Growth hormone abnormal (Investigations) | 1 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 16 (35) | 8 (18)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 8 (16) | 7 (13)
Neutrophil count decreased (Investigations) | 13 (19) | 4 (6)
Platelet count decreased (Investigations) | 19 (42) | 14 (33)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 2 (11)
Weight loss (Investigations) | 3 (3) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 12 (22) | 12 (18)
Blood glucose increased (Metabolism and nutrition disorders) | 16 (33) | 18 (42)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (8) | 4 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (5) | 4 (5)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (8) | 2 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 7 (13) | 9 (14)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 4 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (6)
Abducens nerve disorder (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 6 (7) | 3 (4)
Dysgeusia (Nervous system disorders) | 11 (18) | 4 (7)
Headache (Nervous system disorders) | 6 (8) | 10 (13)
IVth nerve disorder (Nervous system disorders) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 3 (7)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (9)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (13) | 6 (12)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (7)
Depression (Psychiatric disorders) | 1 (1) | 2 (5)
Insomnia (Psychiatric disorders) | 2 (4) | 7 (13)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (4)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (3) | 1 (4)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 17 (35)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (29) | 12 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (20) | 13 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 5 (12) | 4 (7)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 12 (23) | 7 (13)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less